CLINICAL TRIAL: NCT06543771
Title: Clinical Performance Study of Safety Test ABO Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diagast (Industry)
Collaborators: Soladis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPSP_23-07
Record Dates: First submitted 2024-06-19; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Transfusion Reaction
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: In situ used for near patient In vitro Medical device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Safety Test ABO and ABTest Card® — Pre transfusional control with the Safety Test ABO device (reference device) and the ABTest Card® device (comparator).

SUMMARY:
The study aims to confirm the performance equivalence of the in vitro diagnostic device Safety Test ABO with the ABTest Card device.

DETAILED DESCRIPTION:
According to the regulatory text "Common specifications for certain class D in vitro diagnostic medical devices in accordance with Regulation (EU) 2017/746 of the European Parliament and of the Council" [2], 90% of the results will be derived from the performance study carried out at the DIAGAST laboratory on tube left over and blood bag, and 10% of the results will be derived from the use of the device in a real situation ("at the bedside").

Regulation 2017/746 (IVDR) on IVDMD has been effective since May 2022 with transitional periods. The IVDR replaces the current EU Directive (98/79/EC) to ensure a higher level of health and safety for the making available and putting into service of medical devices on the EU market. As the Safety Test ABO and ABTest Card® are already CE marked under Directive 98/79/EC as List IIA product, this study is part of the device's post-marketing performance monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old for the category marked with *.
* Undergo capillary blood sampling;
* Belong to one of the clinical category:

  * Patient in need of blood transfusion without any pathology known to have an impact on transfusion act*;
  * Patient in need of blood transfusion suffering from congenital erythrocyte pathology (sickle cell anaemia, beta thalassemia)*
  * Patient in need of blood transfusion suffering from haematology disease (eg. cancer), or undergoing haemodialysis*;
  * Patient with cold agglutinin*;
  * Premature patient with gestational age < 37 weeks of newborn ≤27 days old in need of blood transfusion;
  * Newborn eligible for Guthrie Test;
  * Newborn eligible for glycemic test.
* Have health care insurance;
* Have given his/her written consent (or legal representative in case of newborn);

Exclusion Criteria:

* Pregnant woman;
* Person deprived of liberty;
* Unconscious person;
* Person under guardianship or trusteeship;
* For neonatal clinical category: age ≥28 days and <18 years old.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Concordance obtained between blood type information from medical record and patient results obtained by Safety Test ABO. | 5 minutes.
  Comparison of the "patient" blood type determined from the results of the Safety Test ABO device (A, B, AB, O) with the "patient" blood type in the medical record (A, B, AB, O).
Concordance obtained between blood bag labelling information and blood bag results obtained by Safety Test ABO. | 5 minutes.
  Comparison of the "donor" blood type determined from the results of the Safety Test ABO device (A, B, AB, O) with the "donor" blood type shown on the blood bag label (A, B, AB, O).
Concordance obtained on patient blood type between Safety Test ABO and ABTest Card® results. | 5 minutes.
  Comparison of the "patient" blood type determined from the results of the ABTest Card® device (A, B, AB, O) with the "patient" blood type determined from the results of the Safety Test ABO device (A, B, AB, O).
Concordance obtained on blood bag blood type between Safety Test ABO and ABTest Card® results. | 5 minutes.
  Comparison of the "donor" blood type determined from the results of the ABTest Card® device (A, B, AB, O) with the "donor" blood type determined from the results of the Safety Test ABO device (A, B, AB, O).
Blood compatibility between blood bag and patient for the Safety Test ABO. | 5 minutes.
  Comparison of the "patient" blood type determined from the results of the Safety Test ABO device (A, B, AB, O) with the "donor" blood type determined from the results of the Safety Test ABO device (A, B, AB, O).
Blood compatibility between blood bag and patient for the ABTest Card®. | 5 minutes.
  Comparison of the "patient" blood type determined from the results of the ABTest Card® device (A, B, AB, O) with the "donor" blood type determined from the results of the ABTest Card® device (A, B, AB, O).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided